CLINICAL TRIAL: NCT05042921
Title: Pediatric Patients With Spinal Muscular Atrophy in China: A Nationwide Registry
Brief Title: Pediatric Spinal Muscular Atrophy (SMA) China Registry
Status: Active, not recruiting | Type: Observational
Sponsor: Biogen (Industry)
Responsible Party: Sponsor
Other Study IDs: CN-SMG-11774
Record Dates: First submitted 2021-09-08; First posted 2021-09-13 (Actual); Last update posted 2025-09-03 (Actual); Status verified 2025-09

CONDITIONS: Muscular Atrophy, Spinal
MeSH Terms: conditions — Muscular Atrophy, Spinal

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 60 Months
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- DMT Treated Participants: Participants with SMA who received prior treatment with DMTs including nusinersen will be followed prospectively for up to 60 months and the available data is collected retrospectively.
- Untreated Participants: Participants with SMA who received no treatment will be followed prospectively for up to 60 months.

SUMMARY:
The primary objective of the study is to describe the natural history and utilization of disease modifying therapy (DMT) treatments among pediatric Chinese participants with spinal muscular atrophy linked to chromosome 5q (5q-SMA). The study will examine SMA natural history and DMT outcomes in a real-world setting both prospectively and retrospectively.

ELIGIBILITY:
Key Inclusion Criteria:

* Ability of the participant and/or his/her legally authorized representative (e.g., parent or legal guardian), as appropriate and applicable, to understand the purpose and risks of the study, to provide informed consent, and to authorize the use of confidential health information in accordance with national and local privacy regulations.
* Genetically confirmed 5q-SMA.
* Age < 18 years at enrollment.

Key Exclusion Criteria:

* Unable or unwilling to provide informed consent.
* Other types of SMA (non 5q-SMA).

NOTE: Other protocol defined inclusion/ exclusion criteria may apply.

Max Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Study Population: Pediatric participants with 5q-SMA will be enrolled to obtain information on both the natural history of the disease and effectiveness and safety of DMTs.
Sampling Method: Probability Sample
Enrollment: 600 (Actual)
Dates: Start 2021-11-18 (Actual); Primary Completion 2027-09-02 (Estimated); Study Completion 2027-09-02 (Estimated)

PRIMARY OUTCOMES:
Natural History and Utilization of Disease Modifying Therapy (DMT) Treatments Among Pediatric Chinese Participants With Spinal Muscular Atrophy Linked to Chromosome 5q (5q-SMA) | Up to 60 months

OTHER OUTCOMES:
Effectiveness of DMT Treatments | Up to 60 months
  Effectiveness will be assessed using following measures: time to mortality, motor function, motor measures, pulmonary function, scoliosis, hospitalizations and comorbidities, clinical observations, patient reported outcomes, wheelchair use, nutrition and electrophysiology and biomarkers.
Safety of DMT Treatments | Up to 60 months
  Safety will be assessed by adverse events (AEs) and serious AEs.

CONTACTS AND LOCATIONS:
Overall Officials: Medical Director, Study Director — Biogen
Locations (25):
- China (25):
  - Anhui Children's Hospital, Hefei, Anhui
  - Beijing Children's Hospital, Capital Medical University, Beijing, Beijing Municipality
  - Children's Hospital of Chongqing Medical University, Chongqing, Chongqing Municipality
  - Fujian Medical University Union Hospital, Fuzhou, Fujian
  - Xiamen Maternal and Child Health Hospital, Xiamen, Fujian
  - The First Affiliated Hospital, Sun Yat-sen University, Guangzhou, Guangdong
  - Shenzhen Children's Hospital, Shenzhen, Guangdong
  - Maternity and Child Health Care of Guangxi Zhuang Autonomous Region, Nanning, Guangxi Zhuang
  - The Second Hospital of Hebei Medical University, Shijiazhuang, Hebei
  - The Third Affiliated Hospital of Zhengzhou University, Zhengzhou, Henan
  - Hunan Children's Hospital, Changsha, Hu'nan
  - Xiangya Hospital, Central South University, Changsha, Hu'nan
  - Wuhan Children's Hospital, Tongji Medical College Huazhong University of Science & Technology, Wuhan, Hubei
  - The Affiliated Hospital of Inner Mongolia Medical University, Hohhot, Inner Mongolia
  - Xuzhou Central Hospital, Xuzhou, Jiangsu
  - Jiangxi Provincial Children's Hospital, Nanchang, Jiangxi
  - The First Hospital of Jilin University, Changchun, Jilin
  - Children's Hospital Affiliated to Shandong University, Jinan, Jinan Shandong
  - Dalian Women and Children's Medical Group, Dalian, Liaoning
  - Shengjing Hospital of China Medical University, Shenyang, Liaoning
  - People's Hospital of Ningxia Hui Autonomous Region, Yinchuan, Ningxia Hui
  - Children's Hospital of Fudan University, Shanghai, Shanghai Municipality
  - The Second Affiliated Hospital of Xi'An Jiaotong University, Xi’an, Shanxi
  - West China Second University Hospital, Sichuan University, Chengdu, Sichuan
  - The Children's Hospital, Zhejiang University School of Medicine, Hangzhou, Zhejiang

IPD SHARING:
Plan to Share IPD: Yes
In accordance with Biogen's Clinical Trial Transparency and Data Sharing Policy on https://www.biogentrialtransparency.com/
URL: https://vivli.org/